CLINICAL TRIAL: NCT03837431
Title: Diagnosis of Cutaneous Leishmaniasis Using the CL-Detect Rapid Test in Ethiopia
Brief Title: Cutaneous Leishmaniasis Diagnostic Study
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 1219/18
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cutaneous Leishmaniases
Keywords: Cutaneous; Leishmaniasis; Ethiopia; RDT
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin samples will be stored (skin slit smear, dental broach sample, tape sample) for a period of one year after the end of the study for quality assurance testing. If patients consented to long-term storage and secondary use of their samples, the skin samples will be stored for a period up to 25 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CL suspicion: Individuals presenting with clinical suspicion of CL
  Interventions: Diagnostic Test: Skin slit; Diagnostic Test: Dental broach; Diagnostic Test: Tape disc

INTERVENTIONS:
Diagnostic Test: Skin slit — Skin slit microscopy, RDT and PCR
Diagnostic Test: Dental broach — Dental broach RDT and PCR
Diagnostic Test: Tape disc — Tape disc PCR

SUMMARY:
The performance of the CL Detect Rapid test will be tested in individuals with suspected cutaneous leishmaniasis in Ethiopia using both skin slit and dental broach samples against a combined reference of microscopy and PCR. Alternative sampling methods will also be evaluated.

DETAILED DESCRIPTION:
Cutaneous Leishmaniasis is common in Ethiopia and mainly affects the poor living in rural areas. Diagnosis of CL routinely uses invasive skin slits which are examined with microscopy, requiring trained staff and an equipped lab. A new rapid diagnostic test for CL which may be used in the field has been developed and validated in several countries where other Leishmania species are present. Less invasive tape sampling has also become available. Whether this new RDT and alternative sampling methods can be used in Ethiopia is unclear.

The performance of the CL detect Rapid Test against a combined reference (microscopy and PCR) and alternative sample collection methods will be tested in CL suspected individuals in North-West Ethiopia in a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

- Clinical suspicion of CL

Exclusion Criteria:

* ≤ 2 years of age
* Not willing or able to provide consent/assent
* CL presentation with only lesions for which skin slit samples cannot be obtained (e.g. eyelids)
* Co-morbidity with visceral leishmaniasis
* On CL treatment at time of enrollment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting at the LRTC with clinically suspected CL during the study period will be screened for eligibility. Suspicion for CL is assessed by physicians as per routine care. In general, children are included in the study population since they are commonly affected, and also make up the majority of DCL patients. Very young children below the age of two are excluded as was done in other studies18 since the study does require more potentially painful procedures as compared to the routine diagnostic procedures.
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity of CL detect Rapid Test using skin slit sampling | February 2019
  % test positive/negative compared against a combined reference of microscopy and PCR with skin slit sampling(positive if any of the two are positive)

SECONDARY OUTCOMES:
Sensitivity, specificity of CL detect Rapid Test using dental broach sampling | February 2019
  CL detect Rapid Test against combined reference of microscopy and PCR using skin slit sampling
Sensitivity, specificity of CL detect Rapid Test with skin slit or dental broach sampling | May 2018
  CL detect Rapid Test with skin slit sample against CL detect Rapid Test with dental broach sample
Sensitivity, specificity of CL detect Rapid Test compared to routine | February 2019
  CL detect Rapid Test positive/negative with skin slit sample compared to microscopy with skin slit sample
Sensitivity, specificity of dental broach sample compared to skin slit sample | February 2019
  PCR with dental broach compared to PCR with skin slit sample
Sensitivity, specificity of tape disc sampling | February 2019
  PCR with tape disc sampling compared to PCR with skin slit sampling
Sensitivity, specificity of routine testing | February 2019
  Microscopy with skin slit sampling compared to PCR with skin slit sampling
Species identification | February 2019
  For selected CL lesions species identification will be done
Immunomodulatory mediators in CL lesions using non-invasive sampling | February 2019
  Tape disc samples will be used and correlation with lesion severity will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Johan van Griensven, MD, PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium; Rezika Mohammed, MD, Principal Investigator — College of Medicine and Health Sciences, University of Gondar, Gondar, Ethiopia
Locations (1):
- Leishmania Research and Treatment Center, University of Gondar hospital, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
IPD accessible by managed access
Supporting Information: Study Protocol
Time Frame: After completion of the primary publication
Access Criteria: Applicants will need to fill out a data access request form
URL: https://www.itg.be/E/data-sharing-open-access

REFERENCES:
- [Derived] van Henten S, Fikre H, Melkamu R, Dessie D, Mekonnen T, Kassa M, Bogale T, Mohammed R, Cnops L, Vogt F, Pareyn M, van Griensven J. Evaluation of the CL Detect Rapid Test in Ethiopian patients suspected for Cutaneous Leishmaniasis. PLoS Negl Trop Dis. 2022 Jan 18;16(1):e0010143. doi: 10.1371/journal.pntd.0010143. eCollection 2022 Jan. PMID 35041672